CLINICAL TRIAL: NCT04165590
Title: Clinical Study of Plasmodium Immunotherapy for Advanced Malignant Solid Tumors
Brief Title: Plasmodium Immunotherapy for Advanced Malignant Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CAS Lamvac Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KGYY-002
Record Dates: First submitted 2019-11-14; First posted 2019-11-18 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Advanced Malignant Solid Tumor
Keywords: advanced malignant solid tumor; Plasmodium immunotherapy; Plasmodiun vivax

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood-stage infection of P.vivax (Experimental): This is a single arm study that is planed to enroll 60 patients with advanced malignant solid tumor and each patient will be vaccinated with P.vivax-infected red blood cells containing approximately 0.1-1.0 × 10^7 Plasmodium parasites. And successful infection will be indicated by microscopic observation of parasitemia in peripheral blood samples. The treatment will last 5-10 weeks from the day of successful infection and will be terminated by antimalarial drugs.
  Interventions: Other: Plasmodium immunotherapy

INTERVENTIONS:
Other: Plasmodium immunotherapy — The patient will be vaccinated with P. vivax-infected red blood cells containing approximately 0.1-1.0 × 10^7 Plasmodium parasites.

SUMMARY:
The purpose of this study is: 1) to evaluate the effectiveness and extended safety of the Plasmodium immunotherapy for the advanced malignant solid tumors. 2) To explore the safe and effective course of the Plasmodium immunotherapy for the advanced malignant solid tumors. 3) To explore the possible indications of Plasmodium immunotherapy for advanced malignant solid tumors.

The treatment will last 5-10 weeks from the day of successful infection and will be terminated by antimalarial drugs.

DETAILED DESCRIPTION:
This study is planed to enroll 60 patients. Each patient will be vaccinated with 2 ml of P. vivax-infected red blood cells, containing approximately 0.1-1.0 × 10^7 Plasmodium parasites. The treatment will last for 5-10 weeks from the day of successful infection. During the period of Plasmodium immunotherapy, doctor will use artesunate to control the P. vivax erythrocyte infection rate at a low level, so as to prevent the severe adverse event. After 5-10 weeks, parasitemia will be terminated by antimalarial drugs for ending the treatment of Plasmodium immunotherapy (the immunological treatment effect may persist after the termination of Plasmodium infection). After the treatment, patients will be followed up for 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-70 years male or female.
2. Patients with advanced maligant solid tumors in lung, liver, prostate, ovary, brain, thyroid and colorectum, etc.
3. Patients with primary central nervous system (CNS) tumor or brain metastases from solid tumors, comply with the following standards can participate in this study: Up to the clinical trial screening period, the imageological examination provides progression-free evidence for at least 3 months, blood brain barrier has not been damaged or is already recovered from the former treatment (surgery or radiotherapy) injury, without intracranial hemorrhage or myelorrhagia history, without metastases to the brain stem, midbrain, pons, medulla oblongata or eye subsidiary organs within 10 mm area (the optic nerve and optic chiasma).
4. The patients have measurable tumors based on the criterion of RECIST1.1.
5. Tumor classification should be determined by histopathology and pathological report should be provided. If tumor tissue is available, before participating in the trail, the research center need to obtain the paraffin blocks or at least 6 unstained sections of the tumor tissue and the relevant pathological reports. If the above tumor tissue samples are not available, samples of any kind (such as fine needle aspiration biopsy samples, cell mass samples (such as pleural, peritoneal effusion samples and lavage samples) are acceptable. If tumor tissue is not available, patients are still eligible for the study.
6. For the patients who previously received one or more of the following therapies, the interval time of the termination of chemotherapy (including interventional chemotherapy) or radiotherapy is at least 28 days for patients who had received chemotherapy or radiotherapy; at least 5 half-life time for patients who had received targeted drug therapy (the half-life of targeted drug is according to the drug instructions).
7. ECGO score is 0 to 2, and euphagia.
8. Expected survival ≥ 3 months.
9. WBC≥3× 10^9/L, PLT ≥ 100× 10^9/L, HGB ≥ 100 g/L, and albumin ≥ 30 g/L, no significant morphological abnormalities of red blood cells, or anemia (iron deficiency anemia, autoimmune hemolytic anemia, thalassemia, etc.).
10. Patients with gastrointestinal bleeding, hemoptysis or other chronic bleeding symptoms were cured before enrollment.
11. Patients with no severe dysfunction of cardiopulmonary, liver and kidney function (child-push grading of liver function A or B, Cr≤ 1.5 x ULN).
12. Patient will be able to understand and sign informed consent.
13. According to the researcher's judgment, the patient's compliance could meet the needs of follow-up.

Exclusion Criteria:

1. Nasopharyngeal cancer, head and neck tumors.
2. HPV positive patients with advanced malignant solid tumors in cervical, anal, vulvar, vaginal and penile.
3. Pancreatic cancer patients.
4. Small cell lung cancer patients.
5. Patients with severe hemoglobin disease or severe G6PD deficiency.
6. Patients with splenectomy or splenomegaly.
7. Patients with drug addiction or alcohol dependence.
8. Have not yet been washed out from the previous therapeutic effects, except the following: the bisphosphonates used for bone metastasis or osteoporosis.
9. Uncontrolled pleural effusion, pericardial effusion or ascites.
10. Tumor-related pain that are uncontrollable.
11. Active malignant tumor metastasis of CNS (progression or controlling the symptoms with anticonvulsants or corticosteroids ).
12. Patients with significant immunodeficiency detection ( CD4+T cell absolute count <200 /ul)
13. With the following diseases or conditions: serious or uncontrolled systemic disease or any unstable systemic diseases (including but not limited to active infection, grade three hypertension, unstable angina, congestive heart failure, class III or IV heart disease, severe arrhythmia, liver and kidney dysfunction or metabolic disease), a clear history of neurological or psychiatric disorders, etc.
14. According to the principal investigator's judgment, any other diseases, metabolic disorders, abnormal results of clinical laboratory tests or physical examination, the diseases that leading to usage of the prohibited drugs, influencing the results reliability, putting patients in high risk.
15. Have undergone major surgery within 4 weeks of the screening period, or plan to undergo major surgery during the study period, PICC catheter and central venous catheter implantation are excluded.
16. Received any antineoplastic drugs, immune cells, antibodies, or vaccines within five drug half-life (not sure the half-life, will be subject to two weeks) during the screening period.
17. Patients who have previously received allogeneic bone marrow transplantation or solid organ transplantation.
18. Receiving any other anti-tumor treatment at the same time.
19. Lung function is seriously damaged, the MNW <39% or can't get out of bed, still feel short of breath when resting.
20. Rough cough, dyspnea, without normal diet or difficult to cooperate.
21. Poor body condition, the researchers assess that the patients can't tolerate the Plasmodium immunotherapy.
22. Pregnant or lactating women.
23. Patients that are unable to comply with the research and follow-up procedure.
24. Any case that the researchers believe that the patient does not suit for this clinical study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-10-24 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 2 years
  Starting from treatment until the disease progression is first found or the time of any cause of death (disease progression refers to tumor growth, or metastasis of primary tumor, or discovery of new lesions).

SECONDARY OUTCOMES:
Tumor marker level | 2 years
  The patient's sensitive tumor markers will be reviewed periodically from the time they are enrolled into the study.
Disease Control Rate | 2 years
  The proportion of patients who had a best response rating of complete response, partial response, or stable disease.
Immunological index | 2 years
  Detection of absolute number of immune cells（such as CD3+CD4+、CD3+CD8+ and so on）in peripheral blood by flow cytometry.
Quality of life score | 2 years
  Patients are regularly filled with QLQ-C30 (cancer patient quality of life scale) to assess the quality of life of the patients.
Overall survival | 2 years
  The time starting from the treatment to death of whatever causes (when subjects have lost for follow-up before death, the last follow-up time will be calculated as the time of death).
1 year of survival rate | 2 years
  The number of cancer cases remaining after 1 year of treatment / the total number of cancer cases treated * 100%.
2 year of survival rate | 2 years
  The number of cancer cases remaining after 2 years of treatment / the total number of cancer cases treated * 100%.
time of tumor progression | 2 years
  TTP is the time between the beginning of treatment and the onset of tumor progression.
Duration of disease control | 2 years
  Duration of disease control is the time from the first evaluation of the tumor as CR, PR or SD to the first evaluation as PD (progressive disease) or any cause of death.
pain score | 2 years
  Patients are regularly evluated with pain assessment scale

CONTACTS AND LOCATIONS:
Overall Officials: Hou Jianghou, Ph.D, Study Director — Yunnan Kungang Hospital
Locations (1):
- Yunnan Kungang Hospital, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chen L, He Z, Qin L, Li Q, Shi X, Zhao S, Chen L, Zhong N, Chen X. Antitumor effect of malaria parasite infection in a murine Lewis lung cancer model through induction of innate and adaptive immunity. PLoS One. 2011;6(9):e24407. doi: 10.1371/journal.pone.0024407. Epub 2011 Sep 9. PMID 21931708
- [Result] Qin L, Chen C, Chen L, Xue R, Ou-Yang M, Zhou C, Zhao S, He Z, Xia Y, He J, Liu P, Zhong N, Chen X. Worldwide malaria incidence and cancer mortality are inversely associated. Infect Agent Cancer. 2017 Feb 14;12:14. doi: 10.1186/s13027-017-0117-x. eCollection 2017. PMID 28228842
- [Result] Yang Y, Liu Q, Lu J, Adah D, Yu S, Zhao S, Yao Y, Qin L, Qin L, Chen X. Exosomes from Plasmodium-infected hosts inhibit tumor angiogenesis in a murine Lewis lung cancer model. Oncogenesis. 2017 Jun 26;6(6):e351. doi: 10.1038/oncsis.2017.52. PMID 28650446
- [Result] Liu Q, Yang Y, Tan X, Tao Z, Adah D, Yu S, Lu J, Zhao S, Qin L, Qin L, Chen X. Plasmodium parasite as an effective hepatocellular carcinoma antigen glypican-3 delivery vector. Oncotarget. 2017 Apr 11;8(15):24785-24796. doi: 10.18632/oncotarget.15806. PMID 28445973
- [Result] Adah D, Yang Y, Liu Q, Gadidasu K, Tao Z, Yu S, Dai L, Li X, Zhao S, Qin L, Qin L, Chen X. Plasmodium infection inhibits the expansion and activation of MDSCs and Tregs in the tumor microenvironment in a murine Lewis lung cancer model. Cell Commun Signal. 2019 Apr 12;17(1):32. doi: 10.1186/s12964-019-0342-6. PMID 30979375
- See also: Free full text. — http://www.ncbi.nlm.nih.gov/pubmed/21931708
- See also: Free full text.This article has been cited by other articles in PMC. — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC5307699/
- See also: Free full text.This article has been cited by other articles in PMC. — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC5519199/
- See also: Free full text. — http://ncbi.nlm.nih.gov/pubmed/28445973
- See also: Free full text. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6461823/